CLINICAL TRIAL: NCT04995380
Title: Validation and Comparison of Scores for Prediction of RIsk for Post-operative Major Morbidity After Cholecystectomy in Acute Calculous Cholecystitis: Protocol for a Prospective Multicenter Observational Study (SPRIMACC)
Brief Title: Validation and Comparison of Scores for Prediction of RIsk for Post-operative Major Morbidity After Cholecystectomy in Acute Calculous Cholecystitis (SPRIMACC)
Acronym: SPRIMACC
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Paola Fugazzola, Medical Doctor, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20210057631
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Early Cholecystectomy — Cholecystectomy performed within 10 days from onset of symptoms

SUMMARY:
The SPRIMACC study is a prospective multicenter observational study with the primary endpoint to prospectively validate the Chole-Risk score in predicting a complicated postoperative course (post-operative major complications (Clavien-Dindo>=3a), length of stay (LOS) > 10 days or need of readmission within 30 days from the discharge) in patients undergoing Early Cholecystectomy (EC) for Acute Calculous Cholecystitis (ACC). The secondary endpoints of the study are to prospectively validate and compare other wellknown risk prediction models (the POSSUM/P-POSSUM score, the Modified Frailty Index (mFI), the Charlson Comorbidity Index (CCI), the American Society of Anesthesiologists (ASA) score and the APACHE II score) in predicting a complicated post-operative course in patients undergoing EC.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of Acute Calculous Cholecystitis (ACC) as defined by Tokyo Guidelines 2018 criteria
* be candidate to Early Cholecystectomy (EC) during the index admission*
* be ≥ 18 years old
* be stratified for the risk of Common Bile Duct Stones (CBDS) according to the Israelian Score, and, in case of confirmation of CBDS receive pre-operative Endoscopic Retrograde Cholangiopancreatography (ERCP).
* provide signed and dated informed consent form
* willing to comply with all study procedures and be available for the duration of the study.

  * All the patients treated with initial open cholecystectomy, those who undergo Early Laparoscopic Cholecystectomy (ELC), those with conversion from laparoscopic to open cholecystectomy or those who undergo bail out procedures (e.g. subtotal cholecystectomy) will be included.

Exclusion Criteria:

* pregnancy or lactation
* acute cholecystitis not related to a gallstone etiology
* onset of symptoms >10 days before cholecystectomy**
* concomitant cholangitis or pancreatitis
* intraoperative treatment of common bile duct stones
* anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

  * Patients with ACC associated with common bile duct stones who underwent pre-operative ERCP could be included if they receive EC within 10 days from onset of symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with ACC as defined according to the Tokyo Guidelines 2018 to one of the participating hospitals will be assessed for eligibility on presentation.
Sampling Method: Probability Sample
Enrollment: 1261 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Complicated post-operative course | 30 days after discharge
  The study outcome is a composite outcome including:
  1. 30-day post-operative major morbidity, intended as Clavien-Dindo >= 3a complication
  2. length of stay (LOS) > 10 days
  3. readmission within 30 days from the discharge
  after Early Cholecystectomy for Acute Calculous Cholecystis. It is a binary outcome (0/1): in the event of a, b or c occurring, the patient's course is defined as complicated (1). If neither a, b, nor c occur, the course is defined as uncomplicated (0).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Fugazzola, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (2):
- Chirurgia 1, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Department of General and Digestive Surgery Hospital Universitario La Princesa, Instituto de Investigación Sanitaria Princesa (IIS-IP) Universidad Autónoma de Madrid (UAM),, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Martino M, Mora-Guzman I, Jodra VV, Dehesa AS, Garcia DM, Ruiz RC, Nisa FG, Moreno FM, Batanero SA, Sampedro JEQ, Cumplido PL, Bravo AA, Rubio-Perez I, Asensio-Gomez L, Aranda FP, Farrarons SS, Moreno CR, Moreno CMM, Lasarte AS, Calvo MP, Aparicio-Sanchez D, Del Pozo EP, Pellino G, Martin-Perez E. How to Predict Postoperative Complications After Early Laparoscopic Cholecystectomy for Acute Cholecystitis: the Chole-Risk Score. J Gastrointest Surg. 2021 Nov;25(11):2814-2822. doi: 10.1007/s11605-021-04956-9. Epub 2021 Feb 24. PMID 33629230
- [Derived] Fugazzola P, Cobianchi L, Di Martino M, Tomasoni M, Dal Mas F, Abu-Zidan FM, Agnoletti V, Ceresoli M, Coccolini F, Di Saverio S, Dominioni T, Fare CN, Frassini S, Gambini G, Leppaniemi A, Maestri M, Martin-Perez E, Moore EE, Musella V, Peitzman AB, de la Hoz Rodriguez A, Sargenti B, Sartelli M, Vigano J, Anderloni A, Biffl W, Catena F, Ansaloni L; S.P.Ri.M.A.C.C. Collaborative Group. Prediction of morbidity and mortality after early cholecystectomy for acute calculous cholecystitis: results of the S.P.Ri.M.A.C.C. study. World J Emerg Surg. 2023 Mar 18;18(1):20. doi: 10.1186/s13017-023-00488-6. PMID 36934276